CLINICAL TRIAL: NCT01531439
Title: Comparison of Two Naloxone Infusion Rates on the Postoperative Recovery of Patients Undergoing Spine Fusion Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Ben J Pieters, Staff Anesthesiologist, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 11 04-059
Record Dates: First submitted 2011-06-20; First posted 2012-02-13 (Estimated); Results first posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Pain, Postoperative; Postoperative Nausea and Vomiting; Scoliosis
Keywords: Narcotic Antagonists; Naloxone infusion; Postoperative pruritis; Patient controlled analgesia; Pediatric; Children
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Scoliosis | interventions — Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naloxone infusion 0.5 mcg/kg/hr (Active Comparator)
  Interventions: Drug: Naloxone
- Naloxone 2.5 mcg/kg/hr (Experimental): Naloxone infusion 2.5 mcg/kg/hr
  Interventions: Drug: Naloxone

INTERVENTIONS:
Drug: Naloxone — Naloxone infusion 0.5 mcg/kg/hr
  Other Names: Narcan
  Arms: Naloxone infusion 0.5 mcg/kg/hr
Drug: Naloxone — Naloxone infusion 2.5 mcg/kg/hr
  Other Names: Narcan
  Arms: Naloxone 2.5 mcg/kg/hr

SUMMARY:
There will be two groups in this study: one group will be given the standard infusion of naloxone, a drug which helps reduce side effects from opioids needed after surgery, and the other group will receive a higher dose. The trial is designed to determine if a higher dose of naloxone infusion will reduce side effects from opioid therapy in patients who have undergone spine fusion for scoliosis.

DETAILED DESCRIPTION:
Currently, patients undergoing spinal fusion for scoliosis are routinely given patient controlled analgesia (PCA) for pain control postoperatively. PCA therapy is typically combined with an ultra low dose naloxone infusion because of the established benefit of reduced pruritis and nausea. The investigators hypothesize that using a higher dose naloxone infusion may lead to further improvement in pruritis and nausea and may improve GI function. Improvement in bowel function could lead to faster initiation of oral intake as well as transition to oral pain medication and even decreased length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic scoliosis requiring spine fusion surgery
* Age 10-21 years

Exclusion Criteria:

* Inability to understand PCA instructions
* Allergy to: morphine, hydromorphone, fentanyl, naloxone, or diphenhydramine
* Chronic opioid therapy > 2 months
* Non-English speaking

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2016-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J. Pieters, DO, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naloxone Infusion 0.5 mcg/kg/hr | Naloxone 2.5 mcg/kg/hr
Started | 41 | 43
Completed | 37 | 42
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naloxone Infusion 0.5 mcg/kg/hr | Naloxone 2.5 mcg/kg/hr | Total
Number analyzed (Participants) | 37 | 42 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37 | 42 | 79
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 37 | 71
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 37 | 41 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Hours Until Tolerating Oral Intake
Description: Defined as time when awakening after surgery until tolerating orals.
Time Frame: Assessed daily in hospital while in hospital until taking orals, average 4 days.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Naloxone Infusion 0.5 mcg/kg/hr | Naloxone 2.5 mcg/kg/hr
Number analyzed (Participants) | 37 | 42
hours | 25.9 [19.4 to 29.8] | 25.0 [18.8 to 28.0]

2. Secondary Outcome: Severity of Itching
Description: Visual analog scale presented to subject to complete daily. Minimum value 0 "none" to maximum value 10 "worst possible". Higher scores represent worse outcome.
  Title of scale "Itching VAS".
  Scores were assessed daily for 5 days and an average of the five days was reported.
Time Frame: Assessed daily while in hospital requiring PCA
Measure: Median (Inter-Quartile Range); unit: score on a scale, averaged
Arm/Group | Naloxone Infusion 0.5 mcg/kg/hr | Naloxone 2.5 mcg/kg/hr
Number analyzed (Participants) | 37 | 42
score on a scale, averaged | 2.1 [0.6 to 3.7] | 1.9 [0.6 to 3.7]

3. Secondary Outcome: Severity of Nausea
Description: Nausea VAS presented to subject daily. Zero minimum "none" to 10 maximum "worse possible". Higher scores represent worse clinical outcome.
  Name of scale "Nausea VAS".
  Scores were assessed daily for 5 days and an average of the five days reported.
Time Frame: Assessed daily while in hospital requiring PCA.
Measure: Median (Inter-Quartile Range); unit: score on a scale, averaged
Arm/Group | Naloxone Infusion 0.5 mcg/kg/hr | Naloxone 2.5 mcg/kg/hr
Number analyzed (Participants) | 37 | 42
score on a scale, averaged | 2.0 [0.5 to 3.2] | 1.2 [0.3 to 2.8]

4. Secondary Outcome: Severity of Pain
Description: Visual analog scale for pain. Zero "none" minimum to 10 "worse possible" maximum.
  Name of scale "Pain VAS".
  Scores were assessed daily for 5 days and an average of the five days was reported.
Time Frame: Assessed by bedside nurse 3 times daily while requiring PCA
Measure: Median (Inter-Quartile Range); unit: units on a scale, averaged
Arm/Group | Naloxone Infusion 0.5 mcg/kg/hr | Naloxone 2.5 mcg/kg/hr
Number analyzed (Participants) | 37 | 42
units on a scale, averaged | 3.7 [2.7 to 5.1] | 4.1 [3.0 to 5.6]

ADVERSE EVENTS:
Arm/Group | Naloxone Infusion 0.5 mcg/kg/hr | Naloxone 2.5 mcg/kg/hr
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/42
Other Adverse Events (participants affected / at risk) | 0/37 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No